CLINICAL TRIAL: NCT06325241
Title: Validating the Use of Frailty Measurements to Predict Care Expectations and Deteriorations in Quality of Life Among People With COPD: A Prospective Cohort Study
Brief Title: Validating the Use of Frailty Measurements to Predict Care & Quality of Life
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Sunita Mulpuru, Staff Physician, Investigator, Ottawa Hospital Research Institute
Other Study IDs: 20200048-01H
Record Dates: First submitted 2023-11-10; First posted 2024-03-22 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Frailty; Care expectations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention. This is an observational study.
  Other Names: there are no other names.

SUMMARY:
The aim of this research program is to validate frailty measurements as a risk stratification tool to predict deteriorations in patient-reported outcomes, to gain a better understanding of patient preferences for care within varying degrees of frailty, and to assess differences in frailty measurement between patients and their clinicians.

This work will provide a foundation in the development of customized interventions for people with COPD and varying degrees of frailty, with the goal of improving quality of life and optimizing health system service delivery for patients and their care givers.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of The Ottawa Hospital Respirology clinic
* Chronic Obstructive Pulmonary Disease diagnosis confirmed by pulmonary function testing.
* English or French speaking

Exclusion Criteria:

* patients with a known diagnosis of severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French or English speaking outpatients of the Ottawa Hospital Respirology clinic who are diagnoses with Chronic Obstructive Pulmonary Disease, which is confirmed by pulmonary function testing who are able to speak on the phone for at least 10 minutes.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory Health Related Quality of Life | 12 months
  measured by the validated short version of St. Georges Respiratory Questionnaire (not a scale).

SECONDARY OUTCOMES:
Burden of symptoms - COPD Assessment | 12 months
  measured with the COPD Assessment Test where 0 means no symptoms and 5 means severe symptoms of COPD.
Burden of symptoms - Dyspnea | 12 months
  measured with the modified Medical Research Council scales. Measured on a scale of 0-4 where 0 means not breathless and 4 is too breathless.
Psycho-social well being - Anxiety | 12 months
  measured with the validated Generalized Anxiety Disorder-7. GAD-7 results vary between 0 and 21, the higher the score, the more anxiety.
Psycho-social well being - Depression | 12 months
  measured with the Patient Health Questionnaire-8 scales. PHQ8 results vary between 0 and 24, where the higher the number, more severe is the persons' level of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT06325241/Prot_SAP_000.pdf
  • Informed Consent Form: Verbal consent (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT06325241/ICF_001.pdf
  • Informed Consent Form: English Information Sheet (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT06325241/ICF_002.pdf